CLINICAL TRIAL: NCT02117817
Title: A Phase I Trial of BKM120 in Combination With Weekly Nabpaclitaxel (Abraxane®) in Patients With Advanced Solid Tumors Followed by a Dose Expansion Phase in Patients With Recurrent Endometrial or Recurrent Ovarian Cancer
Brief Title: Phase I BKM120/Abraxane in Solid Tumors, Expansion Phase Recurrent Endometrial or Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Research cancelled
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101305
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Recurrent Ovarian Cancer; Recurrent Endometrial Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms | interventions — NVP-BKM120; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (BKM120 in Combination with Weekly Nabpaclitaxel) (Experimental)
  Interventions: Drug: BKM120; Drug: Nabpaclitaxel

INTERVENTIONS:
Drug: BKM120
Drug: Nabpaclitaxel — Given IV
  Other Names: Abraxane®

SUMMARY:
The purpose of the first part of this study or the dose escalation portion of the study is to determine what dose of BKM120 and Abraxane is safe to give when the two drugs are used at the same time in patients who are diagnosed with a solid cancer. A solid cancer is a cancer that does not involve the blood, bone marrow or lymph nodes. Dose escalation determines the least toxic and most effect dose of this drug combination for treatment. Once this dose is established, it will be used for the dose expansion phase of the study where we will determine the effect of BKM120 and Abraxane in women diagnosed with a recurrent endometrial or ovarian cancer. We will see whether the combination of both drugs improves the response and survival of patients treated on the two drug regimen. Also we will try to find out whether there are changes in tumors that can help us determine what patients are more likely to respond to BKM120 and Abraxane.

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the safety and tolerability of BKM120 in combination with weekly nabpaclitaxel (Abraxane®) in patients with a recurrent solid tumor and in particular a recurrent endometrial or ovarian cancer.
* To determine the MTD and DLT of BKM120 in combination with weekly nabpaclitaxel (Abraxane®) thereby establishing the recommended phase II dose.

Secondary Objectives:

* Obtain pilot data on the clinical tumor response utilizing RECIST criteria of BKM120 in combination with weekly nabpaclitaxel (Abraxane®) in patients with a history of recurrent endometrial or a recurrent ovarian cancer.
* To determine the progression free survival (PFS) of patients treated with BKM120 and nabpaclitaxel (Abraxane®) and a history of recurrent endometrial or ovarian cancer.
* To explore molecular markers that my serve as potential molecular predictors of response including PIK3CA, mTOR, KRAS, PTEN and p53 mutations as well as amplification of ErbB2.
* To test the predictive value of PIK3CA and KRAS mutations in predicting response to this regimen in women diagnosed with a recurrent endometrial or ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with a recurrent solid tumor in the Phase I portion of the trial or in the Phase II portion of the trial a recurrent endometrial or ovarian cancer, not amenable to treatment by surgery, radiotherapy or chemotherapy.
* ECOG performance status £ 2
* Patients must have at least one site of measurable disease defined by RECIST 1.1 criteria. If the patient has received prior radiation therapy one measurable lesion must be outside the irradiated field. Lesions within an irradiated field will be followed as non-target lesions and considered evaluable. If the only site of measurable disease is within a previously irradiated field then 6 months must have elapsed between the completion of radiation therapy and entry on study to be considered measurable.
* Patients with a recurrent ovarian cancer must have received at least one prior platinum containing regimen.
* Patients diagnosed with a platinum sensitive ovarian cancer may be enrolled if they will no longer benefit from treatment with a platinum agent as determined by their physician or it would be detrimental to treat the patient with a platinum agent due to underlying medical problems.
* Adequate bone marrow function as shown by: ANC ≥ 1.0 x 109/L, Platelets ≥ 100 x 109/L, Hgb > 9 g/dL
* Total calcium (corrected for serum albumin) within normal limits (biphosphonate use for malignant hypercalcemia control is not allowed)
* Magnesium within normal limits for the institution.
* Potassium within normal limits for the institution
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or ≤ 3.0 x upper limit of normal (ULN) if liver metastases are present)
* Serum bilirubin within normal range. For patients with liver metastases, serum bilirubin ≤ 1.5 x ULN. For patients with well documented Gilbert Syndrome total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range. )
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
* Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential defined as sexually mature women who have not undergone a hysterectomy or who have had amenorrhea for at least 12 consecutive months or women who have had six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL.
* Patients with Grade 3 or greater peripheral neuropathy.
* Ability to sign informed consent
* INR ≤ 1.5

Exclusion Criteria:

* Patients who have received prior treatment with a P13K inhibitor.
* Patients who have received prior treatment with Nabplaclitaxel Abraxane®.
* Patients with a known hypersensitivity to BKM120 or to its excipients
* Patients with symptomatic brain metastases are excluded. However, patients with asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior local treatment for CNS metastases > 28 days prior to study entry including radiotherapy or surgery. Patients receiving steroids for CNS metastases may not participate on this study.
* Patients with acute or chronic liver disease, renal disease or pancreatitis
* Patients with the following mood disorders as judged by the Investigator, Sub-Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire:

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or patients with active severe personality disorders (defined according to DSM- IV) are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug.
  * Meets the cut-off score of ≥ 12 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
* Patients with diarrhea ≥ CTCAE 4.0 grade 2
* Patient has active cardiac disease including any of the following:

  * Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO)
  * QTc > 480 msec on screening ECG (using the QTcF formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with document compromise in cardiac function
  * Symptomatic pericarditis
* Patient has a history of cardiac dysfunction including any of the following:

  * Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
* Patient has poorly controlled diabetes mellitus or steroid-induced diabetes mellitus defined as a HgbA1C > 8% or a fasting plasma glucose level > 126 mg/dl.
* Patients without a history of diabetes mellitus need to have a fasting plasma glucose level < 126 mg/dl.
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol

  • Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Please refer to Appendix E for a list of prohibited QT prolonging drugs with risk of Torsades de Pointes. Please recognize that this list may not be all inclusive.
* Patients receiving chronic treatment with steroids or another immunosuppressive agent.

  • Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intr-articular) are allowed.
* Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits.
* Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Appendix B for a list of prohibited inhibitors and inducers of CYP3A. Please recognize that this list may not be all inclusive. (Please note that co-treatment with weak inhibitors of CYP3A is allowed).
* Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must recover to a grade 1 toxicity excluding alopecia before starting the trial
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half- lives prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Double barrier contraceptives must be used through the trial by both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential must have a negative serum pregnancy test ≤ 72 hours prior to initiating treatment.

  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during treatment and for16 additional weeks after stopping treatment... The highly effective contraception is defined as either:

    1. True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    3. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomized male partner should be the sole partner for that patient.
    4. Use of a combination of any two of the following (a+b):

       1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
       2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Oral contraception, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives.
  * Fertile males, defined as all males physiologically capable of conceiving offspring must use condom during treatment and for an additional 16 weeks after stopping treatment.
  * Female partner of male study subject should use highly effective contraception during dosing of any study agent and for 16 weeks after final dose of study therapy.
* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-02-25 (Estimated); Study Completion 2015-02-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | 2 years

SECONDARY OUTCOMES:
Response rate (at the end of the 3 months of therapy) | 2 years
Time to progressive disease | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Darlene Gibbon, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey

IPD SHARING:
Plan to Share IPD: No